CLINICAL TRIAL: NCT02508116
Title: Assessment of Prospective CYP2C19 Genotype Guided Dosing of Anti-Platelet Therapy in Percutaneous Coronary Intervention (ADAPT)
Brief Title: Assessment of Prospective CYP2C19 Genotype Guided Dosing of Anti-Platelet Therapy in Percutaneous Coronary Intervention
Acronym: ADAPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Sony Tuteja, Research Associate, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 820899
Record Dates: First submitted 2015-07-21; First posted 2015-07-24 (Estimated); Results first posted 2018-11-07 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-10

CONDITIONS: Acute Coronary Syndrome; Cardiovascular Diseases
Keywords: pharmacogenetics; clopidogrel; genotype
MeSH Terms: conditions — Acute Coronary Syndrome; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Patients undergoing PCI are randomized to genotype guided antiplatelet therapy vs. usual care.
Oversight: Data Monitoring Committee: No

ARMS (2):
- CYP2C19 Genotype guided (Experimental): Prospective CYP2C19 genotyping to decide antiplatelet therapy.
  Interventions: Genetic: CYP2C19 genotyping
- Control group (No Intervention): Antiplatelet therapy will be decided based on usual care

INTERVENTIONS:
Genetic: CYP2C19 genotyping — The study utilizes a genotyping device, SpartanRx™ (Spartan Bioscience, Ottawa, Canada) that provides identification of a patient's CYP2C19 *2, *3, and *17 genotypes determined from genomic DNA from a buccal swab sample with 1 hour turnaround time
  Other Names: SpartanRx
  Arms: CYP2C19 Genotype guided

SUMMARY:
This is a randomized, prospective, open label study to determine the cost-effectiveness of genotype-guided antiplatelet therapy. Patients undergoing percutaneous intervention (PCI) with stent implantation, will be randomized either to genotype guided dosing of antiplatelet therapy or usual care. The study utilizes a novel genotyping device, SpartanRx, to determine CYP2C19 genotypes from a buccal swab sample with 1 hour turnaround time.

DETAILED DESCRIPTION:
Clopidogrel is a thienopyridine antiplatelet agent, which inhibits the purinergic P2RY12 receptor on platelets and prevents their aggregation. It is commonly used in patients with acute coronary syndromes (ACS) undergoing percutaneous coronary intervention (PCI). CYP2C19 is one of the principal enzymes involved in the bioactivation of clopidogrel from the pro-drug to its active metabolite. The most common loss of function (LOF) allele is *2 (c.681G>A; rs4244285), with frequencies of ~15% in Caucasians and Africans and 29-35% in Asians. A large meta-analysis demonstrated that CYP2C19*2 carriers treated with clopidogrel have a higher risk for major adverse cardiac events compared to noncarriers.Therefore, clopidogrel is less effective in patients who are CYP2C19 poor metabolizers and alternative therapy is recommended. A newer-generation thienopyridine, prasugrel, was found to be associated with a reduction in major adverse cardiac events (death, myocardial infarction, stroke) compared to clopidogrel, but with an increased risk of fatal and major bleeding events.

Now that clopidogrel is available in generic form, pharmacogenetic (PGx) screening could allow for individualized anti-platelet therapy in which patients with functional CYP2C19 alleles could be prescribed clopidogrel, and the more expensive agent would be reserved for patients with poor metabolizer status. A cost-effectiveness analysis of CYP2C19 screening for selection of antiplatelet therapy found that genotype-guided therapy would lead to more cost-effective care rather than uniform usage of either clopidogrel or prasugrel.

A more recent economic evaluation determined that genotyping and prescribing ticagrelor to LOF allele carriers was the most effective strategy when compared against routine clopidogrel or prasugrel use as well as genotyping and prescribing prasugrel to LOF carriers. However, these results were based on decision model of a hypothetical cohort of patients with ACS who underwent PCI and several assumptions were made regarding outcomes, cost and quality of life. True costs associated with genotype guided antiplatelet therapy are unknown. Future prospective studies evaluating the cost effectiveness of a genotype guided approach are needed. We are proposing a pilot study which will provide information necessary for planning a prospective study that will directly estimate events averted, costs, quality-adjust life years (QALYs) and cost per QALY ratios. Information to be obtained in this pilot includes estimates of costs and their variance, preference scores (for calculating QALYs) and their variance, the correlation of cost and effects (required for sample size estimation for cost-effectiveness ratios), event rates, and implementation metrics (to estimate likely penetration of testing in the trial). The results from this study will provide more accurate estimates of the means and variances of cost and QALYs required to plan future trials.

OBJECTIVES

* To identify factors linked with successful implementation of clinical pharmacogenetic (PGx) testing in a large academic medical center.
* To conduct a prospective pilot study to determine means and variances for cost, QALYs and the correlation of cost and effect.
* To determine the rates of clinical outcomes.

APPROACH In the genotype guided arm, a buccal swab will be obtained from subjects immediately following PCI/stent, to determine CYP2C19 genotype with the SpartanRx system. Subject with slow metabolizer status [1 or 2 loss-of-function (LOF) mutations (*2 or *3) in CYP2C19] will be recommended to initiate therapy with prasugrel or ticagrelor in place of clopidogrel. Subjects with normal metabolizer status (homozygous for the *1 allele in CYP2C19) will be recommended to initiate therapy with clopidogrel. Antiplatelet choice is ultimately decided by physician judgment incorporating all clinical factors.

In the control arm, choice of antiplatelet therapy will be decided by treating physician as per usual care. DNA will be collected via a saliva sample to assess CYP2C19 genotype at the conclusion of the study.

Subjects in both groups will complete a baseline health related quality of life questionnaire (HrQoL) and additional clinical data pertaining to cardiac history will be collected from medical records. Subjects will be contacted every three months for medical services utilization, clinical information, and HrQoL assessments for a total of one year.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects, ≥18 to ≤80 years at time of study
2. Status post PCI with stent implantation requiring antiplatelet therapy
3. Willingness to comply with all study-related procedures

Exclusion Criteria:

1. Pending imminent surgery placing patients at increased risk for bleeding with prasugrel or ticagrelor.
2. History of intracranial hemorrhage, TIA, and stroke
3. Active bleeding
4. Need for long-term anticoagulation (i.e. warfarin, dabigatran, rivaroxaban, apixaban, edoxaban, or lovenox).
5. Current or prior (within the past four weeks) treatment with voraxapar (Zontivity).
6. Severe renal or hepatic impairment
7. Treating physician does not want subject to participate
8. Drug allergy to clopidogrel, prasugrel or ticagrelor.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 509 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sony Tuteja, PharmD, MS, Principal Investigator — University of Pennsylvania; Jay S Giri, MD, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Tuteja S, Glick H, Matthai W, Nachamkin I, Nathan A, Monono K, Carcuffe C, Maslowski K, Chang G, Kobayashi T, Anwaruddin S, Hirshfeld J, Wilensky RL, Herrmann HC, Kolansky DM, Rader DJ, Giri J. Prospective CYP2C19 Genotyping to Guide Antiplatelet Therapy Following Percutaneous Coronary Intervention: A Pragmatic Randomized Clinical Trial. Circ Genom Precis Med. 2020 Feb;13(1):e002640. doi: 10.1161/CIRCGEN.119.002640. Epub 2020 Jan 12. PMID 31928229

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients, age ≥18 to ≤80 years at time of study, who were underwent PCI between November 2014 and August 2016 at the Hospital of the University of Pennsylvania or Penn Presbyterian Medical Center.
Period: Overall Study
Arm/Group | CYP2C19 Genotype Guided | Control Group
Started | 252 | 257
Received Intervention as Randomized | 249 | 255
Completed | 244 | 250
Not Completed | 8 | 7
Not completed — Lost to Follow-up | 2 | 3
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Protocol Violation | 1 | 2
Not completed — Physician Decision | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CYP2C19 Genotype Guided | Control Group | Total
Number analyzed (Participants) | 249 | 255 | 504
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (9.7) | 62.9 (10.2) | 62.9 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 66 | 134
  Male | 181 | 189 | 370
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 194 | 197 | 391
  Race: Black | 48 | 51 | 99
  Race: Asian | 6 | 6 | 12
  Race: Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 249 | 255 | 504
Hospital Site [Count of Participants; unit: Participants]
  Hospital of the University of Pennsylvania | 135 | 141 | 276
  Penn Presbyterian Hospital | 114 | 114 | 228
Acute coronary syndrome [Count of Participants; unit: Participants] | 124 | 129 | 253
Insurance Status [Count of Participants; unit: Participants]
  Public | 100 | 110 | 210
  Other | 149 | 145 | 294
Work Status [Count of Participants; unit: Participants]
  Full time | 88 | 92 | 180
  Retired | 84 | 85 | 169
  Disabled | 12 | 13 | 25
  Not provided | 45 | 44 | 89
  Other/unknown | 20 | 21 | 41
Tobacco use [Count of Participants; unit: Participants]
  Never | 114 | 123 | 237
  Former | 105 | 94 | 199
  Current | 28 | 37 | 65
  unknown | 2 | 1 | 3
Medical history [Count of Participants; unit: Participants]
  Hypertension | 190 | 199 | 389
  Hypercholesterolemia | 112 | 113 | 225
  Diabetes Mellitus | 89 | 79 | 168
  Previous MI | 63 | 67 | 130
  Previous PCI | 83 | 83 | 166
  Previous CABG | 32 | 36 | 68
  Previous Stroke | 7 | 15 | 22
P2Y12 inhibitor use prior to admission [Count of Participants; unit: Participants]
  Clopidogrel | 80 | 85 | 165
  Prasugrel | 12 | 9 | 21
  Ticagrelor | 2 | 6 | 8
  None | 155 | 155 | 310
Pharmacotherapy prior to admission [Count of Participants; unit: Participants]
  Aspirin | 165 | 157 | 322
  ACE inhibitor or ARB | 115 | 109 | 224
  Beta-blocker | 121 | 125 | 246
  Calcium channel blocker | 50 | 62 | 112
  Statin | 112 | 113 | 225
  Other anti-anginal | 83 | 78 | 161

OUTCOME MEASURES:

1. Primary Outcome: The Number (Percentage) of Participants Receiving Prasugrel/Ticagrelor
Description: The number (percentage) of participants receiving prasugrel/ticagrelor in each randomized arm
Time Frame: for up to 7 days after PCI
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | CYP2C19 Genotype Guided | Control Group
Number analyzed (Participants) | 249 | 255
Participants
  Clopidogrel | 174 | 201
  Prasugrel/ticagrelor | 75 | 54
Statistical Analysis 1: Comparison: CYP2C19 Genotype Guided vs Control Group; The sample size calculation was based on two factors: 1) the rate of pre-study prasugrel/ticagrelor use (~20%) and 2) anticipated increase in prasugrel/ticagrelor prescribing based on the frequency CYP2C19 LOF variants (~30-35%). We estimated a 15% difference in the use of prasugrel/ticagrelor in the two groups (35% in the genotyped group and 20% in the control group). A sample size of 138 per group (a total of 276) would provide 80% power at an alpha level of 0.05 to detect this difference; Test type: Superiority; p = 0.03, Regression, Logistic; Odds Ratio (OR) = 1.6, 95% CI 2-sided [1.07 to 2.42]

2. Secondary Outcome: Number of Participants With Drug Orders in Agreement With the Genotype-guided Recommendations
Description: Agreement to suggested treatment recommendations based on genotype. The agreement rate was defined as the number of participants in genotyped group with loss of function variants that received prasugrel or ticagrelor + the number of participants without these variants that received clopidogrel divided by the total number in this group.
Time Frame: for up to 7 days after PCI
Population: Subjects with genotype data available
Measure: Count of Participants; unit: Participants
Arm/Group | CYP2C19 Genotype Guided | Control Group
Number analyzed (Participants) | 242 | 226
Participants | 172 | 133

3. Secondary Outcome: Number of Participants With Major Cardiac Events
Description: major cardiac events defined as occurrence of first myocardial infarction, ischemic stroke, cardiovascular death, stent thrombosis, or need for urgent revascularization
Time Frame: 1 year
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | CYP2C19 Genotype Guided | Control Group
Number analyzed (Participants) | 249 | 255
Participants | 34 | 26
Statistical Analysis 1: Comparison: CYP2C19 Genotype Guided vs Control Group; The incidence of first MACE between the groups were compared by use of Kaplan-Meier estimators; statistical tests were based on log-rank tests; Test type: Superiority; p = 0.27, Log Rank

4. Secondary Outcome: Number of Participants With Bleeding Events
Description: major bleeding events defined by the Bleeding Academic Research Consortium (BARC) type 3 or 5.
  Type 3= Overt bleeding requiring: blood transfusion, surgical intervention or intravenous vasoactive agents; cardiac tamponade; intracranial hemorrhage; intraocular bleeding.
  Type 5= fatal bleeding
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | CYP2C19 Genotype Guided | Control Group
Number analyzed (Participants) | 249 | 255
Participants | 6 | 7

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | CYP2C19 Genotype Guided | Control Group
All-Cause Mortality (participants affected / at risk) | 8/249 | 7/255
Serious Adverse Events (participants affected / at risk) | 132/249 | 115/255
Other Adverse Events (participants affected / at risk) | 28/249 | 34/255
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYP2C19 Genotype Guided (N=249) | Control Group (N=255)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
angina pectoris (Cardiac disorders) | 33 (33) | 21 (21)
angina unstable (Cardiac disorders) | 1 (1) | 1 (1)
atrial fibrillation (Cardiac disorders) | 4 (4) | 3 (3)
bradyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
cardiac arrest (Cardiac disorders) | 3 (3) | 0 (0)
cardiac failure (Cardiac disorders) | 2 (2) | 1 (1)
cardiac failure congestive (Cardiac disorders) | 3 (3) | 4 (4)
cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
myocardial infarction (Cardiac disorders) | 8 (8) | 11 (11)
pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
tachyarrhytmia (Cardiac disorders) | 1 (1) | 0 (0)
stent thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 5 (5)
ventricular arrythmia (Cardiac disorders) | 3 (3) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
gastrointestinal hemmorhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
gastrointestinal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
melena (Gastrointestinal disorders) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
rectal hemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
drug intolerance (General disorders) | 1 (1) | 1 (1)
bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
cardiac transplantation (Cardiac disorders) | 0 (0) | 1 (1)
lung transplant rejection (Immune system disorders) | 0 (0) | 1 (1)
bronchitis (Infections and infestations) | 1 (1) | 1 (1)
cellulitis (Infections and infestations) | 0 (0) | 1 (1)
endocarditis (Infections and infestations) | 1 (1) | 1 (1)
gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
groin abscess (Infections and infestations) | 1 (1) | 0 (0)
influenza (Infections and infestations) | 0 (0) | 1 (1)
osteomyelitis (Infections and infestations) | 0 (0) | 2 (2)
pneumonia (Infections and infestations) | 4 (4) | 5 (5)
septic shock (Infections and infestations) | 1 (1) | 0 (0)
coronary artery restenosis (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
subdural hematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
hemoglobin decrease (Investigations) | 1 (1) | 0 (0)
diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
rectal mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
dizziness (Nervous system disorders) | 1 (1) | 0 (0)
epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
ischemic stroke (Nervous system disorders) | 2 (2) | 2 (2)
polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
syncope (Nervous system disorders) | 3 (3) | 0 (0)
transient ischemic attack (Nervous system disorders) | 1 (1) | 0 (0)
confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
acute renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
hematuria (Renal and urinary disorders) | 0 (0) | 2 (2)
renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
angioplasty (Surgical and medical procedures) | 5 (5) | 3 (3)
aortic valve replacement (Surgical and medical procedures) | 3 (3) | 0 (0)
coronary artery bypass grafting (Surgical and medical procedures) | 5 (5) | 3 (3)
gastrectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
implantable defibrillator implantation (Surgical and medical procedures) | 6 (6) | 0 (0)
knee arthroplasty (Surgical and medical procedures) | 3 (3) | 1 (1)
mitral valve repair (Surgical and medical procedures) | 0 (0) | 3 (3)
rotator cuff repair (Surgical and medical procedures) | 1 (1) | 0 (0)
percutaneous coronary intervention (Surgical and medical procedures) | 4 (4) | 2 (2)
aortic aneursym (Vascular disorders) | 1 (1) | 1 (1)
aortic dissection (Vascular disorders) | 0 (0) | 1 (1)
hypotension (Vascular disorders) | 1 (1) | 1 (1)
peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYP2C19 Genotype Guided (N=249) | Control Group (N=255)
angina pectoris (Cardiac disorders) | 6 (6) | 11 (11)
atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
palpitation (Cardiac disorders) | 1 (1) | 0 (0)
vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
hematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
melena (Gastrointestinal disorders) | 0 (0) | 2 (2)
mouth swelling (Gastrointestinal disorders) | 1 (1) | 0 (0)
drug intolerance (General disorders) | 0 (0) | 2 (2)
malaise (General disorders) | 0 (0) | 1 (1)
edema peripheral (Gastrointestinal disorders) | 1 (1) | 0 (0)
abscess (Infections and infestations) | 0 (0) | 1 (1)
urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
upper limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
dizziness (Nervous system disorders) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 0 (0) | 2 (2)
calculus ureteric (Renal and urinary disorders) | 0 (0) | 1 (1)
hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
dyspnea (Reproductive system and breast disorders) | 0 (0) | 3 (3)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
eye hemorrhage (Eye disorders) | 0 (0) | 1 (1)
eye pain (Eye disorders) | 1 (1) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
dental pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
confusional state (Psychiatric disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/16/NCT02508116/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/16/NCT02508116/SAP_001.pdf